CLINICAL TRIAL: NCT06069544
Title: A Randomized, Dose-escalation Phase I/IIa Trial With Controlled Human Malaria Infection to Evaluate Safety, Tolerability, Immunogenicity and Efficacy of an Investigational RNA-based Vaccine for Prevention of P. Falciparum Malaria in Healthy Malaria naïve Adults
Brief Title: A Clinical Trial to Evaluate the Safety, Efficacy and Immune Responses After Vaccination With an Investigational RNA-based Vaccine Against Malaria
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BNT165-02
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Malaria
Keywords: RNA vaccine; Vaccine; Active immunization against malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BNT165e (Experimental): Escalating dose levels
  Interventions: Biological: BNT165e
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT165e — Multi-antigen RNA-based vaccine for active immunization against malaria administered as intramuscular injection
  Arms: BNT165e
Other: Placebo — Isotonic NaCl solution (0.9%)
  Arms: Placebo

SUMMARY:
This is a randomized, dose-escalation Phase I/IIa trial to evaluate safety, tolerability, immunogenicity and efficacy of an investigational RNA-based vaccine (BNT165e) for prevention of P. falciparum malaria in healthy malaria-naive adults.

The multi-antigen malaria vaccine (designated BNT165e) is a combination of three distinct RNAs, BNT165c and BNT165d (composed of BNT165d1 and BNT165d2), encoding P. falciparum antigens encapsulated in lipid nanoparticles. The BNT165c RNA encodes the full Plasmodium falciparum circumsporozoite protein. The BNT165d1 and BNT165d2 RNAs both encode conserved, immunogenic segments of liver stage-expressed proteins.

DETAILED DESCRIPTION:
Part A of this trial will be observer-blind and assess the reactogenicity, safety, and immunogenicity of up to 9 dose combinations in a 3-dose regimen of the 3 components of BNT165e. One dose combination will also be tested in a Day 1, Day 29, and Day 57 dosing schedule in Cohort 10. Participants will be randomized 5:1 active:placebo.

In Cohorts 1 to 9, the initial two doses will be administered ~8 weeks apart and the third dose will be administered ~18 weeks after the second dose. In Cohort 10, the investigational medicinal product (IMP) will be administered 28 days apart on Day 1, Day 29, and Day 57.

Participants who are out of window for dosing in the event of a trial pause can be discontinued from further vaccination. If a participant is discontinued either from further vaccination or discontinued from the trial, the sponsor can decide to replace this participant with a new participant. Participants will be randomized to the vacancy in the open cohort until that cohort has filled. The number of participants may be increased up to 177 in the event of participant replacement or re-enrollment.

The planned trial duration is up to a maximum of 84 weeks for each participant in Cohorts 1 to 9, and 66 weeks for each participant in Cohort 10. Trial duration may exceed the listed maximum time in the event of a trial pause.

An amendment will be submitted to the Health Authorities detailing Part B, which will explore the efficacy of BNT165e in a controlled human malaria infection model.

ELIGIBILITY:
Inclusion Criteria:

* Have given informed consent by signing and dating the informed consent form (ICF) before initiation of any trial-specific procedures.
* Are willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions and other requirements of the trial. This includes that they are able to understand and follow trial-related instructions.
* Are aged 18 to 55 years, have a body mass index over 18.5 kg/m^2 and under 35 kg/m^2 and weigh at least 45 kg at Visit 0.
* Are healthy, in the clinical judgment of the investigator based on volunteer-reported medical history data, and physical examination, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory test outcomes at Visit 0.

  * Note: Healthy volunteers with pre-existing stable disease (e.g., obesity, hypertension), defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 90 days before Visit 0, can be included.
* Agree not to enroll in another trial with an IMP starting from Visit 0 and until 12 weeks after receiving Dose 3.
* Have not traveled and agree not to travel to a malaria-endemic region, as defined per Centers for Disease Control and Prevention (CDC) (https://www.cdc.gov/malaria/travelers/country_table/a.html) starting 6 months before Visit 0 and continuously until 28 days after receiving Dose 3.
* Negative human immunodeficiency virus -1 and -2 blood test result at Visit 0.
* Negative Hepatitis B surface antigen test result at Visit 0 and negative anti-Hepatitis C virus (anti-HCV) antibodies, or negative HCV polymerase chain reaction test result if the anti-HCV is positive at Visit 0.
* Volunteers of childbearing potential (VOCBP) that have a negative serum beta-human chorionic gonadotropin pregnancy test result at Visit 0 and negative urine pregnancy test results before each IMP administration. Volunteers born female who are postmenopausal or permanently sterilized will not be considered VOCBP.
* VOCBP who agree to practice a highly effective form of contraception starting at Visit 0 and continuously until 90 days after receiving Dose 3.
* VOCBP who agree not to donate or cryopreserve eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting at Visit 0 and continuously until 90 days after receiving Dose 3.
* Men who have not had a vasectomy and are sexually active with partners of childbearing potential and who agree to use condoms and to practice a highly effective form of contraception with their sexual partners of childbearing potential during the trial, starting at Visit 0 and continuously until 90 days after receiving Dose 3.
* Men who are willing to refrain from sperm donation, starting at Visit 0 and continuously until 90 days after receiving Dose 3.

Exclusion Criteria:

* History of Plasmodium parasitemia (any species) based on volunteer-reported medical history.
* Prior residence for ≥6 months continuously in a malaria-endemic region as defined per CDC (https://www.cdc.gov/malaria/travelers/country_table/a.html) at any point during their lifetime.
* Breastfeeding or intending to become pregnant or to father children starting with Visit 0 and continuously until 90 days after receiving Dose 3.
* History of any serious adverse reactions to vaccines or to vaccine components such as lipids, and including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had an anaphylactic adverse reaction to pertussis vaccine as a child).
* Current or history of the following medical conditions:

  1. Uncontrolled or moderate or severe respiratory diseases (e.g., asthma, chronic obstructive pulmonary disease); symptoms of asthma severity as defined in the US National Asthma Education and Prevention Program Expert Panel report, 2020 - e.g., exclude a volunteer who:

     * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
     * Uses high dose inhaled corticosteroids (per American Academy of Allergy Asthma and Immunology), or
     * In the past year has either of the following:

       * Greater than one exacerbation of symptoms treated with oral/parenteral corticosteroids
       * Needed hospitalization, or intubation for asthma.
  2. History of Diabetes mellitus type 1 or type 2, including cases controlled with diet alone or elevated hemoglobin A1C ≥6.5% at screening (not excluded: history of isolated gestational diabetes).
  3. Hypertension:

     * If a person has a history of hypertension, or elevated blood pressure detected during screening, exclude for blood pressure that is not well controlled. Well controlled blood pressure is defined as consistently ≤140 mm Hg systolic and ≤90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤150 mm Hg systolic and ≤100 mm Hg diastolic at screening and enrollment.
  4. Malignancy within 5 years of screening, excluding localized basal or squamous cell skin cancer.
  5. Any current or history of cardiovascular diseases, (e.g., myocarditis, pericarditis, myocardial infarction, congestive heart failure, cardiomyopathy or clinically significant arrhythmias), unless such disease is not considered relevant for participation in this trial in the investigator's judgment.
  6. An abnormal screening ECG (i.e., showing the corrected QT interval by Fridericia [QTcF] greater than 450 ms; significant ST-T wave changes suggestive of myocardial ischemia or of an acute or indeterminate-age myocardial infarction; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions; complete right or left bundle branch block [QRS greater than 120 ms]; second-or third-degree atrioventricular block); or other clinically significant abnormalities on the ECG at the investigator's discretion.
  7. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
  8. Seizure disorder: History of seizure(s) within the past 3 years or has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Documented major psychiatric illness, including bipolar disorder, major depressive disorder, schizophrenia, autism, and attention deficit-hyperactivity disorder that at the discretion of the investigator could interfere with participation and follow-up as outlined by the trial.
* The following diseases associated with immune dysregulation:

  * Primary immunodeficiencies.
  * History of solid organ or bone marrow transplantation.
  * Asplenia: any condition resulting in the absence of a functional spleen.
  * Currently existing or history of autoimmune disease including and not limited to thyroid autoimmune disease, multiple sclerosis, psoriasis, etc.
* Previous vaccination with an approved or investigational malaria vaccine at any time or having taken part in a human malaria challenge study.
* Receipt of any investigational product within 28 days before Visit 0.
* Any planned non-trial vaccinations starting at Visit 0 and continuously until 28 days after Dose 3.

  * Note: Seasonal influenza and Coronavirus Disease 2019 (COVID-19) vaccines are allowed; however, they should be administered at least 14 days before or 28 days after any IMP administration. Emergency vaccinations, such as tetanus, are allowed to be administered when medically indicated.
* Received blood/plasma products, monoclonal antibodies or immunoglobulin within 120 days before Visit 1 or planned administration starting at Visit 0 and continuously until the last trial visit (365 days after Dose 3).
* Received allergy treatment with antigen injections within 28 days before and after each IMP administration.
* Current or planned treatment with immunosuppressive therapy, including systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent) starting at Visit 0 and continuously until 28 days after Dose 3. Intraarticular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Have a history of alcohol abuse or drug addiction within 1 year before Visit 0 or have a history (within the past 5 years) of substance abuse, which in the opinion of the investigator, could compromise their wellbeing if they participate as participants in the trial, or that could prevent, limit, or confound the protocol specified assessments.
* Any existing condition which may affect vaccine injection and/or assessment of local reactions at the injection site, e.g., tattoos, severe scars, etc.
* Are vulnerable individuals as per International Council for Harmonisation (ICH) E6 definition, i.e., are individuals whose willingness to volunteer in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.
* Any screening hematology and/or blood chemistry laboratory value (per the US FDA 2007) that meets the definition of a Grade ≥2 abnormality or a Grade 1 abnormality at the investigator's discretion at Visit 0 or a Visit 0 troponin above the reference range. Individuals with abnormal but not clinically significant parameters not included in the toxicity guidance may be considered eligible at discretion of investigator, with the exception of abnormal troponin values.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of solicited local reactions at the injection site (pain, erythema/redness, induration/swelling) recorded up to 7 days after each dose | Up to 7 days after each dose
  For each cohort in participants receiving at least one dose of trial intervention.
Frequency of solicited systemic reactions (vomiting, diarrhea, headache, fatigue, muscle/joint pain, and fever) recorded up to 7 d after each dose | Up to 7 days after each dose
  For each cohort in participants receiving at least one dose of trial intervention.
Frequency of participants with at least one adverse event occurring until 28 days after each dose | Up to 28 days after each dose
  For each cohort in participants receiving at least one dose of trial intervention.
Frequency of participants with at least one medically attended adverse event occurring until 24 weeks after last received IMP dose | Up to 24 weeks after last received IMP dose
  For each cohort in participants receiving at least one dose of trial intervention
Frequency of participants in each cohort with at least one serious adverse event occurring until 24 weeks after last received IMP dose | Up to 24 weeks after last received IMP dose
  For each cohort in participants receiving at least one dose of trial intervention.

SECONDARY OUTCOMES:
Descriptive statistics on antibody levels (including geometric means and 95% confidence interval) at assessed timepoints | Up to 365 days after last received IMP dose
  For each cohort - Anti-CSP immunoglobulin G

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (5):
- United States (5):
  - AMR Tempe, Tempe, Arizona
  - University of Maryland, Center for Vaccine Development, Baltimore, Maryland
  - AMR Las Vegas, Las Vegas, Nevada
  - AMR Knoxville, Knoxville, Tennessee
  - Clinical Trials of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mo AX, McGugan G, Pesce JT. Meeting report: Expert consultation on late arresting replication competent (LARC) malaria sporozoite vaccine research & development. Vaccine. 2025 Apr 30;54:127009. doi: 10.1016/j.vaccine.2025.127009. Epub 2025 Apr 16. PMID 40245769